CLINICAL TRIAL: NCT02166021
Title: Phase 2 Trial to Investigate the Clinical Efficacy & the Optimal Administration (Based on the Immunological, Clinical & Neuroradiological Effects) of Autologous Mesenchymal Bone Marrow Stem Cells in Active & Progressive Multiple Sclerosis
Brief Title: Clinical Efficacy of Autologous Mesenchymal Bone Marrow Stem Cells in Active & Progressive Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dimitrios Karussis (Other)
Responsible Party: Sponsor-Investigator, Dimitrios Karussis, Head of The Center for Multiple Sclerosis & Unit of Neuroimmunology, Hadassah Medical Organization
Organization: Hadassah Medical Organization (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: MSC-MS-001-IL
Record Dates: First submitted 2014-05-20; First posted 2014-06-18 (Estimated); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Multiple Sclerosis (MS)
Keywords: Multiple Sclerosis (MS); Stem Cells
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: Patients were randomised into three groups and treated intrathecally (IT) or intravenously (IV) with autologous MSCs or placebo. At 6-months, treatment groups were crossed over and patients re-treated with either MSC or placebo
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (3):
- IT- Treated (Experimental): Injection to IT (Group 1). After 6 months, 8 patients (group 1A) will be treated with MSC once again in IT, and 8 additional patients (group 1B) will receive a placebo.
  Interventions: Biological: Mesenchymal stem cells
- IV - Treated (Experimental): Injection to IV (Group 2). After 6 months, 8 patients (group 2A) will be treated with MSC once again in IV, and 8 additional patients (group 2B) will receive a placebo.
  Interventions: Biological: Mesenchymal stem cells
- Placebo (Placebo Comparator): Placebo at the first injection (group 3). After 6 months, 8 patients (group 3A) will be treated with MSC in IT, and 8 additional patients (group 3B) will be treated with MSC in IV.
  Interventions: Biological: Mesenchymal stem cells

INTERVENTIONS:
Biological: Mesenchymal stem cells — A culture of purified MSCs was prepared under aseptic conditions, and cultured for 4 weeks, until they reached confluency, and were then harvested. After sterility was confirmed, the cells resuspended in normal saline at a concentration of 10 × 106/mL to 15 × 106/mL.
  Other Names: Autologous MSC

SUMMARY:
The purpose of this study is to evaluate the clinical efficacy and the optimal way of administration of autologous mesenchymal bone marrow stem cells (MSC) compering intravenous injection and intrathecal injection vs. placebo, in active-progressive Multiple Sclerosis patients.

DETAILED DESCRIPTION:
Mesenchymal stem cells (MSC) induce immune-modulatory and neurotrophic effects and were shown to have an acceptable safety profile for clinical applications. We aimed to evaluate the safety and efficacy of MSC transplantation in active progressive MS and investigate possible neuroprotective effects.

Methods: This single-center double-blind crossover trial enrolled 48 patients with progressive MS (expanded disability status scale (EDSS) range: 3.5-6.5, mean: 5.6+/-0.8). Patients were randomised into three groups and treated intrathecally (IT) or intravenously (IV) with autologous MSCs (1x106/Kg) or placebo. At 6-months, treatment groups were crossed over and patients re-treated with either MSC or placebo. During the 2-months run-in period and the 12-months after treatment, participants were followed using EDSS, 25-foot timed walking, 9-hole peg test, neurocognitive tests, quantitative magnetic resonance imaging (MRI), functional MRI, optic coherence tomography (OCT), visual evoked potentials (VEP), and dynamic visual tests.

ELIGIBILITY:
Inclusion Criteria:

1. Consenting patients fulfilling the Poser's clinical criteria for definite MS
2. Age: 18-65, males and females
3. Duration of disease: >3 years
4. Progressive form of MS: PPMS, SPMS (with/without relapses)
5. EDSS score of 3.5 - 6.5
6. Failure to currently available, registered - first and second line immunomodulatory treatments (at least one).
7. Evidence for new activity of MS during the 3 months before the injection of MSC.

Exclusion Criteria:

1. Patients who were treated with cytotoxic medications during the last 3 months prior to the inclusion.
2. Patients suffering from significant cardiac, renal or hepatic failure or any other disease that may risk the patient or interfere with the ability to interpret the results
3. Patients with active infections
4. Patients with severe cognitive decline or inability to understand and sign the informed consent
5. Patients who received any cellular treatment in the past

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-01-29 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-12-24 (Actual)

PRIMARY OUTCOMES:
Safety Assessment | 6 months for each treatment cycle; the two cycles (each of 6 months duration) will be combined together and provide a single measurement for each group
  The proportions of the patients in the three treatment-groups (MSC-IV, MSC-IT and placebo) who experienced any adverse event.
Neurological efficacy | 6 months for each treatment cycle; the two cycles (each of 6 months duration) will be combined together and provide a single measurement for each group
  The proportions of the patients with treatment failure (increase of the EDSS by 1 point for patients with baseline values of 5.0 or less and of 0.5 degree for baseline EDSS of more than 5.0), confirmed by two consecutive evaluations, in the three treatment-groups.

SECONDARY OUTCOMES:
EDSS score | 6 months for each treatment cycle; the two cycles (each of 6 months duration) will be combined together and provide a single measurement for each group
  Change from baseline to 6 months visit post each treatment cycle in EDSS following treatment with intravenous or intrathecal MSC infusion, vs. placebo treatment in MS patients at 6 months post treatment. [A decrease in EDSS indicates clinical improvement].
Ambulation score | 6 months for each treatment cycle; the two cycles (each of 6 months duration) will be combined together and provide a single measurement for each group
  Change from baseline to 6 months visit post each treatment cycle in ambulation score following treatment with intravenous or intrathecal MSC infusion, vs. placebo treatment in MS patients at 6 months post treatment. [A decrease in ambulation score indicates clinical improvement].
Functional scores | 6 months for each treatment cycle; the two cycles (each of 6 months duration) will be combined together and provide a single measurement for each group
  Change from baseline to 6 months visit post each treatment cycle in the sum of all functional scores (from the EDSS scoring) following treatment with intravenous or intrathecal MSC infusion, vs. placebo treatment in MS patients at 6 months post treatment. [A decrease in the sum of functional scores indicates clinical improvement].
Single injection vs. repeated MSCs injection | 12 months: ie the total duration of the trial
  Change from baseline to final 12-month visit, in EDSS following treatment of a single injection of MSCs vs. repeated MSCs injections treatment. [A decrease in EDSS indicates clinical improvement].
  *similar comparison will be performed for the ambulation score and the sum of all functional systems' scores
Relapse rate | 12 months: ie the total duration of the trial
  Annualized MS-Relapse rate during the 6 months of each treatment cycle, in the three treatment groups.
T2-weighted flair lesions load in MRI | 6 months for each treatment cycle; the two cycles (each of 6 months duration) will be combined together and provide a single measurement for each group
  The annualized rate of change in the total lesions load of the T2-weighted MRI scans during the 6 months of each cycle of treatment versus the rate of change in the run-in period (before the treatment). [An increase in the volume of lesions indicates progression of the disease].
Total brain volume in MRI | 6 months for each treatment cycle; the two cycles (each of 6 months duration) will be combined together and provide a single measurement for each group
  The annualized rate of change in total brain volume in MRI scans during the 6 months of each cycle of treatment versus the rate of change in the run-in period (before the treatment). [A decrease in the brain volume indicates progression of the disease].
Gadolinium enhancing lesions in MRI | 6 months for each treatment cycle; the two cycles (each of 6 months duration) will be combined together and provide a single measurement for each group
  The mean annualized number of gadolinium-enhancing lesions during the 6 months of each treatment cycle, in the three treatment groups. [The appearance of gadolinium-enhancing lesions in MRI indicates activity of the disease].
Functional MRI | 6 months for each treatment cycle; the two cycles (each of 6 months duration) will be combined together and provide a single measurement for each group
  The annualized rate of change in the z-scores of the motor networks in resting functional MRI during the 6 months of each cycle of treatment versus the rate of change in the run-in period (before the treatment). [An increase in the z-score indicates functional improvement].
  * similar measurements will apply for the pyramidal and visual networks
25-feet timed walking | 6 months for each treatment cycle; the two cycles (each of 6 months duration) will be combined together and provide a single measurement for each group
  The mean time to walk 25-feet during the 6 months in each treatment cycle vs the mean time during the run-in pre-treatment period. [A decrease in the value of timed walking indicates clinical improvement].
9-hole peg test | 6 months for each treatment cycle; the two cycles (each of 6 months duration) will be combined together and provide a single measurement for each group
  The mean time to perform the 9-hole peg test of hands dexterity during the 6 months in each treatment cycle vs the mean time during the run-in pre-treatment period. [A decrease in the value of timed walking indicates clinical improvement].
Paced Auditory Serial Addition Test (PASAT) | 6 months for each treatment cycle; the two cycles (each of 6 months duration) will be combined together and provide a single measurement for each group
  The score given in this neuropsychological test reflects the assess capacity and rate of information processing and sustained and divided attention. This perform during the 6 months in each treatment cycle vs the mean time during the run-in pre-treatment period. [An increase in z score indicates clinical improvement]
Cognitive function: Controlled Oral Word Association Test (COWAT) | 6 months for each treatment cycle; the two cycles (each of 6 months duration) will be combined together and provide a single measurement for each group
  The annualized rate of change in the z-scores of the COWAT cognitive test during the 6 months of each cycle of treatment versus the rate of change in the run-in period (before the treatment). [An increase in the z-score indicates functional improvement].
  * similar measurements will apply for other cognitive tests (SDMT)
Optical coherence tomography (OCT) | 6 months for each treatment cycle; the two cycles (each of 6 months duration) will be combined together and provide a single measurement for each group
  Change from baseline to 6 months visit, post each treatment cycle retinal nerve fiber layer (RNFL) thickness in OCT, following treatment with intravenous or intrathecal MSC infusion, vs. placebo treatment in MS patients at 6 months post treatment. [An increase in RNFL thickness indicates clinical improvement].
  * similar measurements will apply for Macula thickness
Immunology | 6 months for each treatment cycle; the two cycles (each of 6 months duration) will be combined together and provide a single measurement for each group
  Change from baseline to 6 months visit post each treatment cycle in the proportion of the lymphocytes expressing the CD4+CD25+ markers (T-regulatory cells) following treatment with intravenous or intrathecal MSC infusion, vs. placebo treatment at 6 months post treatment. [An increase in the proportion may indicate beneficial effects].
  * similar measurements (for evaluation of safety of the treatment) will be performed for additional white blood cell subpopulations

CONTACTS AND LOCATIONS:
Overall Officials: Hadas Lemberg, PhD, Study Chair — Director, R&D Division
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Derived] Petrou P, Kassis I, Ginzberg A, Hallimi M, Karussis D. Effects of Mesenchymal Stem Cell Transplantation on Cerebrospinal Fluid Biomarkers in Progressive Multiple Sclerosis. Stem Cells Transl Med. 2022 Mar 3;11(1):55-58. doi: 10.1093/stcltm/szab017. PMID 35641166
- [Derived] Petrou P, Kassis I, Levin N, Paul F, Backner Y, Benoliel T, Oertel FC, Scheel M, Hallimi M, Yaghmour N, Hur TB, Ginzberg A, Levy Y, Abramsky O, Karussis D. Beneficial effects of autologous mesenchymal stem cell transplantation in active progressive multiple sclerosis. Brain. 2020 Dec 1;143(12):3574-3588. doi: 10.1093/brain/awaa333. PMID 33253391